CLINICAL TRIAL: NCT07011628
Title: Transition to Ambulatory Bariatric Surgery (TABS) Trial
Acronym: TABS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jason Samuels, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250548
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Obesity-related Medical Conditions; Bariatric Surgery
Keywords: ambulatory surgery; same day discharge; gastric bypass; sleeve gastrectomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same Day Discharge (Active Comparator): Patients in the same day discharge will be discharged from the hospital following surgery without an overnight stay in the hospital.
  Interventions: Other: Same Day Discharge
- Standard of care - Hospital Admission (No Intervention): Patients in the standard of care arm will be admitted to the hospital for at least one overnight stay in the hospital.

INTERVENTIONS:
Other: Same Day Discharge — Patients in the same day discharge arm will be discharged from the hospital within 6 hours of arriving to the recovery unit and without an overnight stay in the hospital.
  Arms: Same Day Discharge

SUMMARY:
This study will compare same day discharge and at least one night stay in the hospital after bariatric surgery. Patients undergoing bariatric surgery will be randomized (i.e. have an equal chance of either plan) to either group. The study's primary outcome is the frequency patients in the study require a visit to the emergency room within 7 days of their surgery.

DETAILED DESCRIPTION:
This pragmatic, parallel, randomized, open-label trial aims to determine the safety and feasibility of same day discharge (SDD) for bariatric surgery including sleeve gastrectomy and gastric bypass. Investigators will investigate the frequency of 7-day emergency department visits with SDD after bariatric surgery (Aim 1). In addition, the investigators will compare total 30-day charges between participants who undergo same day discharge versus those receive post-operative hospital admission (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 60 kg/m2
* Primary Sleeve gastrectomy or Gastric Bypass,
* Undergoing bariatric surgery at sponsor site

Exclusion Criteria:

* Type 1 Diabetes
* Myocardial Infarction
* Unstable Angina or Heart Failure
* Prior Stroke
* Solid organ transplantation
* Systemic glucocorticoid prior 28 days
* Severe Obstructive Sleep Apnea
* Uncontrolled Hypertension (Systolic > 150, Diastolic > 90)
* Untreated Hyperthyroidism
* Chronic Kidney Disease (EGFR < 60)
* Current anticoagulant use,
* Poorly controlled Type 2 diabetes (Hemoglobin A1c in last 3 months > 8.5%)
* Chronic opioid use
* Insulin dependence.
* Need for extended venous thromboembolic event prophylaxis,
* > 1 lifetime bariatric surgery (revisional or conversion bariatric surgery)
* Patient lives > 130 miles from the hospital.
* Tobacco use in last 12 months
* Desire to become pregnant or active pregnancy
* Prisoners
* Unable or unwilling to follow-up
* Unable to understand or provide consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Emergency Department Visits | baseline to seven days
  Number of emergency room visits after surgery

SECONDARY OUTCOMES:
Readmissions to the hospital | baseline to 30 days
  Study personnel will investigate the incidence of readmissions to the hospital in the post-surgical period.
The number of operations or procedures | baseline to 30 days
  Study personnel will compare the frequency of reoperations and procedural interventions after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All participant-level data will be preserved and shared. Shared data will be deidentified prior to sharing. Clinicaltrials.gov will document recruitment progress and final results. Study protocols will be shared with publications as supplementary data and made available upon request. All participant consent document will be collected and stored electronically utilizing the REDCap study data repository. The REDCap data warehouse will also contain the study data dictionary. Study protocols have also been published on the ClinicalTrials.gov and any protocol amendments will be reflected on the ClinicalTrials.gov study page. The investigators will utilize the Research Electronic Data Capture (REDCap) data warehouse maintained locally at Vanderbilt for all data collection. Upon study completion and prior to closing the REDCap data warehouse for this study, the investigators will archive all data after removing patient identifiers in the Open Science Framework data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Per institutional policy, data will be maintained in the local REDCap data repository for 6 years after closure of the study. Following this period, data will be deidentified and uploaded to the OSF repository, which has funding for at least 50 years of data storage.
Access Criteria: Data will be made available upon request after completion of appropriate institutional review board approval and data use agreement obtainment.